CLINICAL TRIAL: NCT01837329
Title: A Phase I Study of Tetrathiomolybdate (TM) in Combination With Carboplatin and Pemetrexed in Chemo-Naive Metastatic or Recurrent Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Phase I Study of Tetrathiomolybdate in Combination With Carboplatin/Pemetrexed in Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Megan Baumgart, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46356
Record Dates: First submitted 2013-02-28; First posted 2013-04-23 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Squamous; NSCLC; Adenocarcinoma; Lung Cancer; Tetrathiomolybdate; Copper; Carboplatin; Pemetrexed Platinum; Newly Diagnosed; Chemo-naive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Lung Neoplasms | interventions — tetrathiomolybdate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tetrathiomolybdate (Experimental): Dose Escalation - It is aimed at determining the maximum tolerated dose of TM in combination with carboplatin and pemetrexed.
  Dose Expansion - The dose expansion portion of the study will begin after completion of the dose escalation phase.
  Interventions: Drug: Tetrathiomolybdate

INTERVENTIONS:
Drug: Tetrathiomolybdate — Dose Escalation - Dose level -1: 20 mg TM orally 3 x daily x 21 days in combination with carboplatin IV area under the curve (AUC) = 6 and pemetrexed IV 500/mgm2 day 1 x 1 cycle.
  Dose level 1: 40 mg TM orally 3 x daily x 21 days in combination with carboplatin IV AUC = 6 and pemetrexed IV 500 mg/m2 day 1 x 1 cycle.
  Dose level 2: 60 mg TM orally 3 x daily x 21 days in combination with carboplatin IV AUC = 6 and pemetrexed IV 500 mg/m2 day 1 x 1 cycle.
  Patients in the dose-expansion cohort will continue on carboplatin and pemetrexed (without TM) at the discretion of the treating physician.
  Dose Expansion - Maximum tolerated dose of TM determined from the dose-escalation cohorts combined with carboplatin IV AUC = 6 and pemetrexed IV 500 mg/m2 day 1 x 4 cycles.
  Other Names: TM

SUMMARY:
The main objective of this study is to determine recommended phase II dose and safety of tetrathiomolybdate (TM) in combination with carboplatin and pemetrexed in chemo-naive metastatic or recurrent non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
Platinum resistance is a major limitation in the treatment of advanced non-small cell lung cancer. Previous studies suggest that reduced tumor platinum levels may significantly contribute to platinum resistance and thus poor outcome following platinum-based chemotherapy in lung cancer.

Tetrathiomolybdate (TM) is a fast-acting copper chelator that has been under significant investigation as an anti-cancer strategy due to its anti-angiogenic property. Furthermore, more recent preclinical evidence suggests that combining TM with platinum drugs resulted in higher intratumoral platinum concentration and greater tumor response. The oncologists at the University of Rochester are studying addition of TM to commonly used 1st line platinum-based doublet, carboplatin/pemetrexed, in patients with non-squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

>18 years old Performance status 0-1 Newly diagnosed stage IV non-squamous non-small cell lung cancer or recurrent disease after prior surgery and/or irradiation Patients must not have received prior chemotherapy for any stage non small cell lung cancer Brain metastases allowed provided they have been controlled for ≥ 2 weeks after completion of treatment and remain asymptomatic while off corticosteroids for at least 1 day Patient or primary care taker must be informed of and understand the investigational nature of this study and must sign and give written approved informed consent in accordance with institutional guidelines.

If patient is of childbearing potential, she or he must agree to practice an effective method of birth control prior to study entry, for the duration of study participation, and for 30 days after the last study dose.

Patient has adequate organ functions: serum bilirubin ≤ 2.0 mg/dL; alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN), or ALT ≤ 5 x ULN if the patient has hepatic metastasis; serum creatinine ≤ 1.5 mg/dL or a calculated creatinine clearance of at least 60 mL/min.

Patient has adequate bone marrow reserve: absolute neutrophil count ≥ 1,500, platelet count ≥ 100,000, and hemoglobin ≥ 9.0.

Exclusion Criteria:

Patient receiving any concurrent chemotherapy Patients who received platinum-based chemotherapy for any purpose Patients who had gastric bypass surgery Patients taking copper supplementation for medical reasons Medical and/or psychiatric problems of sufficient severity to limit full compliance with the study or expose patients to undue risk Patients with active and uncontrolled infection Patients with concomitant active malignancy requiring treatment with cytotoxic chemotherapy or radiation therapy (ongoing hormonal therapy for treatment of malignancy would not exclude patients from this trial) Known anaphylactic or severe hypersensitivity to study drugs or their analogs. Patient has failed to recover from any prior surgery within 4 weeks of study entry.

Patient has clinical evidence of copper deficiency (i.e. ceruloplasmin level was less than 15 mg/dL or free serum copper level less than 2.2 g/dL).

Patients with tumors that are epidermal growth factor receptor (EGFR) mutation and anaplastic lymphoma receptor tyrosine kinase (ALK) positive. If biopsy specimen is insufficient or inadequate for EGFR and/or ALK testing, subjects are eligible for the study.

Patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of Safety and Tolerability | 3 years
  Determine phase II dose and safety of TM in combination with carboplatin and pemetrexed in chemo-naive metastatic or recurrent non-squamous non-small cell lung cancer.

SECONDARY OUTCOMES:
Percentage of participants with Complete Response or Partial Response | 3 years
  Determine efficacy of carboplatin and pemetrexed doublet in combination with TM in chemo-naive metastatic or recurrent non-small cell lung cancer.
Time from date of enrollment to disease progression or death | 3 years
Expression of copper transporter by immunohistochemistry | 3 years
  Determine if pretreatment expression of copper transporter by immunohistochemistry predicts clinical outcome following platinum-based chemotherapy in combination with TM
Platinum sensitivity and copper status | 3 years
  Determine if ceruloplasmin level (a surrogate marker for copper status) is associated with platinum sensitivity
Platinum induced toxicity and copper status | 3 years
  Determine if ceruloplasmin level is associated with platinum-induced toxicity.
Impact on blood mineral levels. | 3 years
  To determine if Tetrathiomolybdate affects serum copper, iron, total iron binding capacity, ferritin or zinc levels when combined with platinum-based chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: David Dougherty, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided